CLINICAL TRIAL: NCT07090005
Title: Comparing the Efficacy and Safety of the EndoZipTM System and Apollo Endoscopic Sleeve Gastroplasty (ESG), Followed by Behavioral Modifications, in Obese Patients Who Have Not Achieved Weight Reduction Through Non-surgical Methods.
Brief Title: Comparing the Efficacy and Safety of the EndoZip System and Apollo ESG in Obese Patients
Acronym: ESG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nitinotes Surgical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL00020
Record Dates: First submitted 2025-07-20; First posted 2025-07-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: The EndoZip system is a single-use device, designed to create multiple internal gastric segmentations in the stomach using an endoscopic approach. The device is intended to be used in adult patients with obesity who have a body mass index (BMI) of 30-40 50 kg/m2 and who have not been able to lose weight or maintain weight loss through more conservative measures. The system uses an automated a minimally invasive approach to form wall-to-wall longitudinal attachments anterior and posterior stomach walls, creating multiple plications within.
Who Masked: Participant, Care Provider
Masking Description: Dietitians and medical staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EndoZip System (Experimental): The EndoZip System is a single-use automated suturing device, designed to create multiple internal gastric segmentations in the stomach using an endoscopic approach.
  Interventions: Device: EndoZip System
- OverStitch Endoscopic Suturing System (Active Comparator): Description: The OverStitch ESG is suturing device, designed to create manual suturing in the stomach using an endoscopic approach.
  Interventions: Device: OverStitch Endoscopic Suturing System (ESG)

INTERVENTIONS:
Device: EndoZip System — The EndoZip System is a single-use automated suturing device, designed to create multiple internal gastric segmentations in the stomach using an endoscopic approach.
  Arms: EndoZip System
Device: OverStitch Endoscopic Suturing System (ESG) — The OverStitch ESG is suturing device, designed to create manual suturing in the stomach using an endoscopic approach.
  Arms: OverStitch Endoscopic Suturing System

SUMMARY:
evaluation of the EndoZip system procedure compared to the Apollo ESG procedure in obese patients.

DETAILED DESCRIPTION:
randomized, multicenter, prospective, two-arms, blinded, clinical study will include up to 184 patients (up to 30 patients per site), aimed at evaluating the safety and effectiveness of the EndoZip system procedure, compared to the Apollo ESG procedure, in obese patients who failed to reduce weight with non-surgical weight-loss methods.

Patients will be enrolled at up to 10 clinical sites in US and Europe. Patients who meet the eligibility criteria will be follow up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65
2. BMI ≥ 30 and ≤50 kg/m².
3. Willingness to comply with the substantial behavioral modifications and dietary restrictions as required by the procedure.
4. History of failure with non-surgical weight-loss methods.
5. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, completing IWQOL questionnaire and completing the medically supervised diet and behavior modification program.
6. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits.
7. Ability to give informed consent.
8. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods.
9. *** There will be a quota for at least a) 46 patients with hypertension treated with 2 or more antihypertensive medications and are well control at least 6 months prior to study enrollment , b) 46 patients with type II diabetes mellitus on oral agents only with HgbA1c ≤ 9 at least 6 months prior to study enrollment, excluding Insulin-dependent. Thus the cohort of 184 patients will be stratified into four groups (Obesity, Obesity & HTN, Obesity & DM, obesity &HTN &DM) and block randomized.

Exclusion Criteria:

1. History of foregut or gastrointestinal (GI) surgery (except uncomplicated cholecystectomy or appendectomy)
2. Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions.
3. Prior open or laparoscopic bariatric surgery.
4. Prior surgery of any kind on the esophagus, stomach or any type of hiatal hernia surgery.
5. Any inflammatory disease of the gastrointestinal tract including esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
6. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
7. A gastric mass or gastric polyps > 1 cm in size.
8. A hiatal hernia > 4cm of axial displacement of the z-line above the diaphragm or severe or intractable gastro-esophageal reflux symptoms.
9. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the endoscope.
10. Achalasia or any other severe esophageal motility disorder
11. Severe coagulopathy (INR >1.5) or on anticoagulation therapy.
12. Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months or a HgbA1C ≥ > 9.
13. Diabetics who are treated with GLP-1 and have lost 5% or more of their weight (%TBWL ≥ 5%).
14. Patients who discontinued GLP-1 therapy and regained less than 80% of the weight they had lost prior to starting GLP-1 treatment and within 3 months of discontinued GLP-1 therapy.
15. Patients with any serious health condition unrelated to their weight that would increase the risk of endoscopy
16. Chronic abdominal pain
17. Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation
18. Hepatic insufficiency or cirrhosis
19. Use of an intragastric device prior to this study due to the increased thickness of the stomach wall preventing effective suturing.
20. Active psychological issues preventing participation in a life-style modification program as determined by a psychologist
21. Patients unwilling to participate in an established medically supervised diet and behavior modification program, with routine medical follow-up.
22. Patients receiving daily prescribed treatment with high dose aspirin (> 80mg daily), anti-inflammatory agents, anticoagulants or other gastric irritants.
23. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication
24. Patients who are pregnant or breast-feeding.
25. Patients with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs
26. Patients taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti- arrhythmic medications
27. Patients who are taking corticosteroids, immunosuppressants, and narcotics
28. Patients who are taking diet pills
29. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
30. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
31. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma) or immunocompromised.
32. Specific diagnosed genetic disorder such as Prader Willi syndrome.
33. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
34. Known history of endocrine disorders affecting weight such as uncontrolled hypothyroidism.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean percent of total body weight loss (%TBWL) after 12 months in Group A patients versus Group B. | 12 months
Percentage of patients in Group A with a reduction in %TBWL of at least 5% at 12 months | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Lenox Hill Hospital | Northwell Health, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided